CLINICAL TRIAL: NCT03635203
Title: C-shaped Root Canal System Prevalence and Configurations of Mandibular First and Second Molars in an Egyptian Sub-population Evaluated by Cone-beam Computed Tomography: A Cross-Sectional Observational Study
Brief Title: C-shaped Root Canal Prevalence and Configurations in Egyptians
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Abdel Aziz, Master student at Endodontic department. Faculty of Oral and Dental Medicine, Cairo University
Other Study IDs: C-shaped_root_canal
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: C-shaped Root Canal
Keywords: C-shaped root canal / C-shaped canals
MeSH Terms: interventions — Cone-Beam Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — A total of 374 CBCT scans of mandibular first and second permanent molars belonging to Egyptian individuals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: CBCT — Observation of C-shaped root canal in mandibular first and second molars in Egyptian sub-population
  Other Names: Cone beam computed tomography

SUMMARY:
The aim of this study is to investigate the prevalence and configuration of C-shaped root canal of mandibular first and second molars among members of an Egyptian sub-population using cone beam computed tomography (CBCT). The prevalence and distribution of the C-shape canal configurations with respect to gender and age will be also investigated.

Data regarding the prevalence and configurations of C-shaped root canal in the first and the second mandibular molars in Egyptian sub-population is lacking which might affect the correct implementation of chemo-mechanical instrumentation and obturation.

DETAILED DESCRIPTION:
1. Scientific Background:

   The main goal of conventional root canal treatment is to prevent or heal apical periodontitis through cleaning, shaping and three-dimensional obturation of the root canal system. To establish this goal; recognition of root canal anatomy is required to minimize the risk of treatment failure.

   Studies recorded variations among different ethnicities in the prevalence and configurations of some root canal systems in particular interest is the root canal configurations of the mandibular first and second molars. Anatomical variations recorded include radix entomolaris, radix paramolaris and C-shaped canal. The prevalence of C-shaped root canal ranges between 2.6% to 44.5% among different ethnicities with the highest percentage in Asian populations.

   C-shaped root canal anatomy has challenges in the diagnosis and endodontic management. Challenge in diagnosis is attributed to the variations in the root canal anatomy that may extend along the entire length of the canal. Preoperative identification of C-shaped root canal and its configurations is difficult by conventional radiographic techniques due to their inherent limitations. Challenges in endodontic management are attributed to the presence of complex isthmi, fins and webs connecting the individual root canals that may complicate the proper cleaning and shaping of the root canal rendering it more difficult. Therefore, it is important to detect and identify the configuration of C-shaped canals before root canal treatment.

   Preoperative recognition of the prevalence and root canal configurations will direct the attention of endodontists to its presence and will facilitate the root canal accessing, negotiation, determining the best three-dimensional instrumentation and obturation technique.
2. Rationale of the study:

Different methods have been used to investigate the prevalence and configurations of C-shaped root canal including: microscopic examination of extracted demineralized teeth after black ink infiltration or microscopic examination for polyester cast resin of the pulp space of demineralized extracted teeth or microscopic examination of extracted teeth with methylene blue dye infiltration followed by resin imbibition, conventional radiography, medical CT and most recently CBCT.

CBCT was reported to be accurate for various root canals morphological analysis because of the 3-dimensional reconstruction of the internal and external morphology of the tooth and high spatial resolution in all planes. It has the ability to investigate the morphology of the root canal system without intervention. Compared to medical CT, CBCT can be accomplished with a substantially lower effective dose and reduced acquisition time.

According to my knowledge, there is only one study that has investigated the prevalence of the C-shaped root canal in mandibular first and second molars among members of sub-Egyptian population, but the configurations of C-shaped root canal have not been studied yet.

Knowledge of the prevalence rate and root canal configurations will direct the attention of endodontists to its presence and will facilitate the root canal accessing, negotiation, determining the best instrumentation and obturation technique thus, long term success rate of the endodontic therapy.

ELIGIBILITY:
Inclusion Criteria:

* CBCT images of good quality at which the mandibular first and second molars could be seen adequately.
* Mandibular first and second molars with fully developed roots.

Exclusion Criteria:

* Tomographic images of poor quality or artifacts interfering with the detection of the root canals
* Tomographic images without demographic data including gender and age of the patient
* Mandibular first and second molars having:
* coronal fillings or deep caries reaching the pulp floor
* root caries specially reaching the bifurcation area or root fracture
* external or internal root resorption
* root canal calcification or a periapical lesion (s)
* previous root canal treatment
* post or crown restoration
* evidence of apicectomy or periapical surgery.
* developmental anomalies.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. The data collection will be obtained from the data base available at a private radiographic center (oral and maxillofacial imaging center located in Cairo, Egypt).
  2. CBCT images will be obtained from Egyptian patients who had CBCT examination as part of their dental examination including diagnosis, treatment planning and follow-up during the years before 2015.
Sampling Method: Probability Sample
Enrollment: 374 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of C-shaped root canal in the whole sample | Immediately
  Using CBCT / Binary system (Yes/No)

SECONDARY OUTCOMES:
Configurations of C-shaped canals of mandibular first and second molars in the whole sample | Immediately
  Using CBCT / Percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan B, Cheung GS, Fan M, Gutmann JL, Fan W. C-shaped canal system in mandibular second molars: Part II--Radiographic features. J Endod. 2004 Dec;30(12):904-8. doi: 10.1097/01.don.0000136206.73115.93. PMID 15564875
- [Background] Fan B, Cheung GS, Fan M, Gutmann JL, Bian Z. C-shaped canal system in mandibular second molars: Part I--Anatomical features. J Endod. 2004 Dec;30(12):899-903. doi: 10.1097/01.don.0000136207.12204.e4. PMID 15564874